CLINICAL TRIAL: NCT03870763
Title: A Randomized, Double-Blind, Double-Dummy, Placebo-Controlled, 3-Arm, Parallel Group Study in Pediatric Subjects Aged 10 Through 17 Years to Evaluate the Efficacy and Safety of BG00012 and BIIB017 for the Treatment of Relapsing-Remitting Multiple Sclerosis
Brief Title: Study to Evaluate the Efficacy and Safety of Dimethyl Fumarate (Tecfidera) and Peginterferon Beta-1a (Plegridy) for the Treatment of Relapsing-Remitting Multiple Sclerosis in Pediatric Participants
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Decision to stop the trial was based on long-term difficulties in fulfilling our enrolment commitments and changes in paediatric MS landscape which no longer support placebo-controlled trials.Decision to stop study was not based on safety concerns.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 800MS301; 2018-000516-22 (EudraCT Number)
Record Dates: First submitted 2019-03-07; First posted 2019-03-12 (Actual); Results first posted 2023-05-16 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Pediatric, Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Dimethyl Fumarate; peginterferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dimethyl Fumarate 240 mg (Experimental): Participants will receive dimethyl fumarate 240 milligrams (mg) capsule twice daily (BID) orally and placebo subcutaneous (SC) injection every 2 weeks for up to 96 weeks (2 years).
  Interventions: Drug: Dimethyl Fumarate
- Peginterferon Beta-1a 125 µg (Experimental): Participants will receive peginterferon beta-1a 125 micrograms (µg) SC injection every 2 weeks and placebo capsule BID orally for up to 96 weeks (2 years).
  Interventions: Drug: Peginterferon Beta-1a
- Placebo (Placebo Comparator): Participants will receive placebo SC injection every 2 weeks and placebo capsule BID orally for up to 96 weeks (2 years)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dimethyl Fumarate — Administered as specified in the treatment arm.
  Other Names: Tecfidera; BG00012
  Arms: Dimethyl Fumarate 240 mg
Drug: Peginterferon Beta-1a — Administered as specified in the treatment arm.
  Other Names: Plegridy; BIIB017
  Arms: Peginterferon Beta-1a 125 µg
Drug: Placebo — Administered as specified in the treatment arm.
  Arms: Placebo

SUMMARY:
The main objective of the study is to evaluate the efficacy of dimethyl fumarate (Tecfidera) and peginterferon beta-1a (Plegridy), both compared with placebo, in pediatric participants with RRMS. The other objectives of this study are to evaluate the safety and tolerability of dimethyl fumarate and peginterferon beta-1a and to assess the effect of dimethyl fumarate and peginterferon beta-1a, both compared with placebo, on additional clinical and radiological measures of disease activity.

DETAILED DESCRIPTION:
Participants will be randomized in a 1:2:2 ratio to receive the double-blind study treatment (Dimethyl Fumarate, Peginterferon Beta-1a, and placebo). Participants experiencing a confirmed relapse or disability progression or high lesion burden on MRI will have the option to discontinue the blinded study treatment and switch to an alternative therapy or open-label BG00012.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a diagnosis of RRMS as defined by the revised consensus definition for pediatric MS
* Must have an EDSS score between 0.0 and 5.0.
* Must have a body weight of ≥30 kg
* Must have experienced ≥1 relapse in the 12 months prior to randomization (Day 1), or must have evidence of asymptomatic disease activity seen on MRI in the 6 months prior to randomization, or ≥2 relapses in the 24 months prior to randomization (Day 1). Relapse is defined as the occurrence of a clinical demyelination event regardless of whether the event is a first or subsequent demyelinating event.

Key Exclusion Criteria:

* Participants having primary progressive, secondary progressive, or progressive RMS.
* Disorders mimicking MS, such as other demyelinating disorders, systemic autoimmune disorders, metabolic disorders, and infectious disorders.
* History of clinically significant cardiovascular, pulmonary, GI, hepatic, renal, endocrinologic, hematologic, immunologic, metabolic, dermatologic, growth, developmental, psychiatric (including depression), neurologic (other than MS), and/or other major disease and/or laboratory abnormality indicative thereof, that would preclude participation in a clinical study
* Occurrence of an MS relapse within the 30 days prior to randomization (Day 1) and/or the subject has not stabilized from a previous relapse prior to randomization

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (23):
- Research Site, Raleigh, North Carolina, United States
- Research Site, Medellín, Colombia
- Research Site, Tallinn, Estonia
- Research Site, Budapest, Hungary
- Research Site, Ar Ramtha, Jordan
- Malaysia (2):
  - Research Site, Petaling Jaya
  - Research Site, Seberang Jaya
- Mexico (3):
  - Research Site, Guadalajara
  - Research Site, Morelia
  - Research Site, Santa Cruz
- Saudi Arabia (2):
  - Research Site, Dammam
  - Research Site, Riyadh
- Research Site, Seoul, South Korea
- Taiwan (2):
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Research Site, Bangkok, Thailand
- Tunisia (4):
  - Research Site, Manouba
  - Research Site, Monastir
  - Research Site, Sfax
  - Research Site, Tunis
- Turkey (Türkiye) (3):
  - Research Site, Ankara
  - Research Site, Izmir
  - Research Site, Samsun

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at the investigative sites in Estonia, Tunisia, Turkey, Jordan and Taiwan from 19 March 2019 to 21 July 2022.
Pre-assignment Details: A total of 11 participants were enrolled and treated in this study.
Groups:
- Dimethyl Fumarate 240 mg: Participants received dimethyl fumarate 120 milligrams (mg) capsules twice daily (BID), orally for 7 days followed by 240 mg capsules, BID, orally for 95 weeks and peginterferon beta-1a matching placebo subcutaneous (SC) injection once every 2 weeks (Q2W) for up to 96 weeks.
- Peginterferon Beta-1a 125 µg: Participants received peginterferon beta-1a, 63 micrograms (µg) on Day 1, 94 µg at Week 2, 125 µg SC injection Q2W from Week 4 up to 96 weeks and peginterferon beta-1a matching placebo SC injection, Q2W for up to 96 weeks.
- Placebo: Participants received peginterferon beta-1a matching placebo SC injection Q2W and dimethyl fumarate matching placebo capsules BID, orally for up to 96 weeks.
Period: Overall Study
Arm/Group | Dimethyl Fumarate 240 mg | Peginterferon Beta-1a 125 µg | Placebo
Started | 2 | 6 | 3
Completed | 2 | 3 | 2
Not Completed | 0 | 3 | 1
Not completed — Study terminated by sponsor | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Worsening of multiple sclerosis attack | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who had received at least 1 dose of study treatment.
Groups:
- Dimethyl Fumarate 240 mg: Participants received dimethyl fumarate 120 mg capsules BID, orally for 7 days followed by 240 mg capsules, BID, orally for 95 weeks and peginterferon beta-1a matching placebo SC injection Q2W for up to 96 weeks.
- Peginterferon Beta-1a 125 µg: Participants received peginterferon beta-1a, 63 µg on Day 1, 94 µg at Week 2, 125 µg SC injection Q2W from Week 4 up to 96 weeks and peginterferon beta-1a matching placebo SC injection, Q2W for up to 96 weeks.
- Total: Total of all reporting groups
Arm/Group | Dimethyl Fumarate 240 mg | Peginterferon Beta-1a 125 µg | Placebo | Total
Number analyzed (Participants) | 2 | 6 | 3 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.5 (2.12) | 15.7 (1.51) | 15.7 (1.15) | 15.6 (1.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 2 | 8
  Male | 1 | 1 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 6 | 3 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 5 | 3 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to First Relapse
Description: A clinical relapse is defined as new or recurrent neurological symptoms, not associated with fever, lasting for at least 24 hours, and followed by a period of 30 days of stability or improvement. Time to relapse is defined as from the first dose of the study drug to the day of relapse. Time to First Relapse is estimated by Kaplan Mayer method.
Time Frame: Baseline up to Week 96
Population: ITT population included all participants who were randomized and received at least 1 dose of study treatment (BG00012, BIIB017, or placebo).
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Dimethyl Fumarate 240 mg | Peginterferon Beta-1a 125 µg | Placebo
Number analyzed (Participants) | 2 | 6 | 3
Days | 413 [413 to 413] | NA [NA to NA] — NA signifies data is not available as no participant in this arm group had a relapse. | 166.5 [113 to 220]

2. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; Initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline up to Week 100
Population: Safety population included all participants who had received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dimethyl Fumarate 240 mg | Peginterferon Beta-1a 125 µg | Placebo
Number analyzed (Participants) | 2 | 6 | 3
Participants
  AEs | 2 | 6 | 3
  SAEs | 1 | 0 | 1

3. Secondary Outcome: Number of New or Newly Enlarging T2 Hyperintense Lesions on Brain Magnetic Resonance Imaging (MRI) Scans at Weeks 48 and 96
Description: The number of new or newly enlarging T2 hyperintense lesions that developed in each participant assessed on magnetic resonance imaging (MRI) scans.
Time Frame: Weeks 48 and 96
Population: ITT population included all participants who were randomized and received at least 1 dose of study treatment (BG00012, BIIB017, or placebo). The overall number of participants analyzed signifies number of participants analyzed in this endpoint and the number analyzed signifies number of participants analyzed at a given timepoint.
Measure: Mean (Full Range); unit: number of lesions
Arm/Group | Dimethyl Fumarate 240 mg | Peginterferon Beta-1a 125 µg | Placebo
Number analyzed (Participants) | 2 | 5 | 3
number of lesions
  Week 48 | 0.5 [0 to 1] | 1.0 [0 to 3] | 3.3 [2 to 4]
  Week 96: number analyzed (Participants) | 2 | 4 | 2
  Week 96 | 2.5 [0 to 5] | 1.3 [0 to 3] | 3.5 [2 to 5]

4. Secondary Outcome: Number of Galdolinium (Gd)-Enhancing Lesions at Weeks 48 and 96
Description: The number of Gd-enhancing lesions was assessed by using MRI scans.
Time Frame: Weeks 48 and 96
Population: as for outcome 3
Measure: Mean (Full Range); unit: number of lesions
Arm/Group | Dimethyl Fumarate 240 mg | Peginterferon Beta-1a 125 µg | Placebo
Number analyzed (Participants) | 2 | 5 | 2
number of lesions
  Week 48 | 0 [0 to 0] | 0 [0 to 0] | 1.5 [0 to 3]
  Week 96: number analyzed (Participants) | 2 | 4 | 2
  Week 96 | 0 [0 to 0] | 0.25 [0 to 1] | 0.5 [0 to 1]

5. Secondary Outcome: Annualized Relapse Rate
Description: A clinical relapse was defined as new or recurrent neurological symptoms, not associated with fever, lasting for at least 24 hours, and followed by a period of 30 days of stability or improvement. The relapse rate for an individual participant was calculated as the number of relapses for that participant divided by the number of participant-years followed. The ARR for each enrolment group was calculated as the total number of relapses experienced in the group divided by the total number of participant-years on the study. An unadjusted relapse rate is reported.
Time Frame: Up to Week 96
Population: as for outcome 1
Measure: Number; unit: relapses per participant year
Arm/Group | Dimethyl Fumarate 240 mg | Peginterferon Beta-1a 125 µg | Placebo
Number analyzed (Participants) | 2 | 6 | 3
relapses per participant year | 0.26 | 0.00 | 0.46

ADVERSE EVENTS:
Time Frame: Baseline up to Week 100
Description: Safety population included all participants who had received at least 1 dose of study treatment.
Arm/Group | Dimethyl Fumarate 240 mg | Peginterferon Beta-1a 125 µg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/6 | 1/3
Other Adverse Events (participants affected / at risk) | 2/2 | 6/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dimethyl Fumarate 240 mg (N=2) | Peginterferon Beta-1a 125 µg (N=6) | Placebo (N=3)
Multiple sclerosis relapse (Nervous system disorders) | 1 | 0 (0) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dimethyl Fumarate 240 mg (N=2) | Peginterferon Beta-1a 125 µg (N=6) | Placebo (N=3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 1
Feeling cold (General disorders) | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 0
Injection site bruising (General disorders) | 0 | 1 | 0
Injection site erythema (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Asymptomatic COVID-19 (Infections and infestations) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Vaginal infection (Infections and infestations) | 1 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 1
Parasite stool test positive (Investigations) | 0 | 1 | 0
Vitamin D decreased (Investigations) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 4 | 1
Multiple sclerosis relapse (Nervous system disorders) | 1 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Sensitive skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated because of long-term difficulties in fulfilling the enrolment commitments and changes in paediatric MS landscape which no longer support placebo-controlled trials. Decision to stop study was not based on safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for non-commercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2019-11-06): https://cdn.clinicaltrials.gov/large-docs/63/NCT03870763/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT03870763/SAP_001.pdf